CLINICAL TRIAL: NCT01392534
Title: Evaluation of the Real-life Efficacy and Safety of a Fixed-dose Telmisartan/Hydrochlorothiazide, Including Its Effect on Plasma Potassium and on Glucose and Lipid Metabolism Parameters in Patients With Essential Arterial Hypertension
Brief Title: Effects of Telmisartan/Hydrochlorothiazide Treatment in Hypertensive Patients Under Real-life Setting
Acronym: POTASSIUM
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Medical Director, Bayer Sp. z o.o. , Poland
Other Study IDs: 15297; KL1010PL (Other: Company Internal)
Record Dates: First submitted 2011-05-26; First posted 2011-07-12 (Estimated); Last update posted 2012-07-04 (Estimated); Status verified 2012-07

CONDITIONS: Primary Hypertension
Keywords: Hypertension; Telmisartan; Hydrochlorothiazide; Potassium; Glucose metabolism; Lipid metabolism
MeSH Terms: conditions — Essential Hypertension; Hypertension | interventions — Telmisartan; Hydrochlorothiazide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Telmisartan/hydrochlorothiazide (Pritor Plus, BAY98-7103)

INTERVENTIONS:
Drug: Telmisartan/hydrochlorothiazide (Pritor Plus, BAY98-7103) — Patients treated with telmisartan/hydrochlorothiazide tablets under the real-life setting. Dosing regimen customised to the needs of each participating patient according to the investigators assessment

SUMMARY:
One of the most common adverse effects resulting from the therapy with thiazides, thiazide-like diuretics and loop diuretics is increased potassium secretion. Disregulation of plasma potassium may be a life-threatening condition due to increased risk of arrythmias. Moreover, it has been postulated that decrease in plasma potassium level may negatively affect glucose metabolism resulting in the increased risk of new-onset type 2 diabetes.The main goal of this study is to assess the efficacy and safety of telmisartan/hydrochlorothiazide in a broad population of hypertensive patients, including the effects of the therapy on plasma potassium level and also on selected parameters of glucose and lipid metabolism.

ELIGIBILITY:
Inclusion Criteria:

* primary hypertension
* age>18 years

Exclusion Criteria:

* Cholestatic disorders or severe hepatic/renal failure
* allergy to telmisartan or hydrochlorothiazide
* treatment-resistant hypokalemia or hypercalcemia
* pregnancy and lactation period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic hypertensive patients not treated with telmisartan/hydrochlorothiazide for approx. 3 mths.
Sampling Method: Probability Sample
Enrollment: 1586 (Actual)
Dates: Start 2010-07; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Change in systolic (SBP) and diastolic (DBP) blood pressure between first and final visit | approx. 3 mths after telmisartan/hydrochlorothiazide treatment initiation

SECONDARY OUTCOMES:
Change in plasma potassium between initial and final visit | approx 3 mths after telmisartan/hydrochlorothiazide treatment initiation
Change in fasting plasma glucose between initial and final visit | approx 3 mths after telmisartan/hydrochlorothiazide treatment initiation
Change in glycated haemoglobin A1C between initial and final visit | approx 3 mths after telmisartan/hydrochlorothiazide treatment initiation
Change in plasma high density lipoprotein between initial and (continued) | approx 3 mths after telmisartan/hydrochlorothiazide treatment initiation
Change in plasma low density lipoprotein between initial and final visit | approx 3 mths after telmisartan/hydrochlorothiazide treatment initiation
Change in plasma cholesterol between initial and final visit | approx 3 mths after telmisartan/hydrochlorothiazide treatment initiation
Change in plasma triglycerides between initial and final visit | approx 3 mths after telmisartan/hydrochlorothiazide treatment initiation
Adverse events collection | approx 3 mths after telmisartan/hydrochlorothiazide treatment initiation

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, Poland